CLINICAL TRIAL: NCT06254638
Title: Effectiveness of a Multicomponent Intervention to Promote Physical Activity Levels During the School Day (MOVESCHOOL)
Acronym: MOVESCHOOL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Extremadura (Other)
Collaborators: Ministry of Science and Innovation, Spain (Other Government)
Responsible Party: Principal Investigator, David Sanchez Oliva, Assistant professor, University of Extremadura
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CNS2022-135604; PID2022-137450OA-I00 (Other Grant/Funding Number: The Spanish Ministry of Science, Innovation and Universities)
Record Dates: First submitted 2024-01-31; First posted 2024-02-12 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Physical Activity; Adolescents; Physical Fitness; Cognition
Keywords: Active Break; Physically active learning; Active Recess; Motivational variables; Sedentary time; Academic indicators
MeSH Terms: conditions — Motor Activity; Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multicomponent school-based intervention (Experimental): The multicomponent intervention will be composed of:
  Physically Active Learning: consists of incorporating physical activity (usually of moderate-vigorous intensity) into the educational content taught in non-physical education academic classes.
  Active breaks: consists of short breaks during non-physical education academic classes that include moderate to vigorous intensity physical activity.
  Active Recess: consists of promoting PA during school breaks. To this end, three strategies will be developed: i) modification of the environment; ii) loose equipment; iii) structured recess. The modification of the environment will consist of providing students with a greater number of spaces for them to be active during recess. Access to sports equipment consists of providing sports equipment to encourage PA practice during recess. Structured recess includes the organization of sports competitions and teacher-led activities.
  Interventions: Behavioral: Multicomponent school-based intervention.
- Control Group (No Intervention): The control group will receive the usual academic classes without any methodological modification during the intervention period.

INTERVENTIONS:
Behavioral: Multicomponent school-based intervention. — Physically active learning: this type of intervention is carried out once a week for 1 hour outside the classroom. The teachers of the corresponding subject (with the support of the research team) are in charge of the physically active classes.
  Active break: the intervention consists of 2 active pauses per day. The development of each pause is carried out through a specific digital platform in which students follow the instructions of an avatar, who is in charge of guiding the realization of the active break. Each active break takes a total of 4 minutes, in which two sets of 20 seconds of work and 10 seconds of rest of four different exercises are performed.
  Active break: The intervention consists of a daily active break, every school day of the week. The design and supervision of each active break will be carried out by the support technician and the teaching staff based on the students' tastes.
  Arms: Multicomponent school-based intervention

SUMMARY:
Study based a multicomponent school-based intervention during the school-day (i.e., Physically active learning, active breaks, and active recess) on Physical Activity, health, educational, and cognition outcomes in adolescents.

DETAILED DESCRIPTION:
MOVESCHOOLS is a quasi-experimental study coordinated by fully qualified researchers in physical activity and sport sciences from two universities [University of Cadiz (UCA) and University of Extremadura (UEX), Spain]. This study is aimed at year 1 to year 3 from Secondary Education students (11-16 years old), belonging to 10 schools in Spain (5 schools in Cadiz and 5 schools in Caceres). The schools will be assigned to a control group (n = 5 schools and 400 students) and an intervention group (n = 5 schools and 400 students). The intervention will last 6 months, and will consist of three components:

1. Inclusion of a physically active classes per week.
2. Development of two daily active breaks of 5 minutes duration.
3. Implementation of daily active recesses.

Before and after the intervention, Physical Activity and sedentary time will be assessed by accelerometry, health-related fitness levels by field tests, body composition parameters by anthropometry, academic performance by school grades, positive health (quality of life and self-perception of health) by questionnaire, and cognitive parameters (executive functions and mathematical fluency) by specific cognition tests. In weeks 8 and 16, Physical Activity and sedentary time will also be evaluated as intermediate measures.

At the end of the intervention the researchers will determine the changes of the main outcome variables. Likewise, the main hypotheses raised will be:

1. Students belonging to the experimental group will improve physical activity and will decrease sedentary time during the school-day when comparing to the students belonging to the control group.
2. Students belonging to the experimental group will result in improved in physical and psychological health markers when comparing to the students belonging to the control group.
3. Students belonging to the experimental group will result in improved academic indicators and cognitive markers when comparing to the students belonging to the control group.
4. Students belonging to the experimental group will improve school climate and motivational variables in academic classes compared to students belonging to the control group.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents in 1st, 2nd and 3rd year of ESO.
* Adolescents with informed consent signed by the family/guardian.
* Schools with at least 80 students enrolled in 1st, 2nd and 3rd ESO.
* Schools belonging to the regions of Cáceres and Cádiz.

Exclusion Criteria:

* Adolescents with any physical disability or health condition that may limit physical activity levels.
* Schools participating in any other physical activity or health promotion program.

Ages: 11 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 900 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Physical activity and sedentary time | 6 months
  Physical activity and sedentary time will be measured through accelerometry (Actigraph GT3X+, Inc., Pensacola, FL, USA).

SECONDARY OUTCOMES:
Cardiorespiratory capacity | 6 months
  The 20-metres shuttle run test will be used to assess cardiorespiratory fitness. Participants will run the 20-metre distance to the rhythm of a recording. The initial speed is 8.5 km/h and will be increased by 0.5 km/h per section. The race will end when the participant stops due to fatigue or when he/she fails to cross the marked lines to the rhythm of the acoustic signals on two consecutive occasions. The last stage or half stage completed by the competitor will be scored.
Musculoskeletal capacity of upper body | 6 months
  The hand grip test will be used to assess musculoskeletal capacity of upper body. The test shall be performed twice with each hand alternately. The maximum score of each hand in kilograms shall be recorded and the mean value between them shall be calculated.
Musculoskeletal capacity of lower body | 6 months
  Standing broad jump shall be used to assess the musculoskeletal capacity of the lower limbs. The participant shall stand behind a line with feet shoulder width apart. The participant is then asked to jump forward as far as possible with both feet. If he/she rests his/her hands or lifts his/her feet off the ground when landing, the test is invalid. The test shall be performed twice, and the best score recorded in centimetres.
Body mass index | 6 months
  Weight and height will be combined to report BMI in kg/m^2.
Body composition | 6 months
  Waist circumference shall be measured as a body composition variable with a non-elastic tape placed in the frontal plane at the midpoint between the upper iliac spine and the costal border at the mid-axillary line. The measurement shall be taken twice and the mean of the two measurements shall be recorded.
Self-reported screen time | 6 months
  Self-reported screen time will be assessed using the Youth Leisure-time Sedentary Behaviour Questionnaire (YLSBQ). Five questions will be selected from the original questionnaire and participants will be asked to answer them by selecting the amount of time they spend per day on each question, ranging from 0 minutes to 5 or more hours.
Subjective physical fitness | 6 months
  The International Fitness Scale will be used for the assessment of subjective physical fitness. Participants will be asked to rate each of the fitness components on a 5-point Likert-type scale ranging from: "very poor" (1); "poor" (2); "fair" (3); "good" (4) and "very good".
Health status | 6 months
  The EuroQol five dimensions three levels will be used to assessment of health status (EQ-5D-3L).This questionnaire is composed of the dimensions of: (i) mobility; (ii) self-care; (iii) usual activities; (iv) pain/discomfort and (v) anxiety/depression. The three levels that participants should mark a Likert-type scale correspond to (i) no problem; (ii) some problems; (iii) many problem.
Self-perceived health | 6 months
  Self-perceived health will be measured through the classic self-reported health item, where participants will have to classify their health among the following options: "excellent" (5); "very good" (4); "good" (3); "fair" (2) and "poor" (1).
School engagement | 6 months
  The engagement scale (UWES-S-9) will be used to evaluate school engagement. The UWES-S-9 is composed of nine items that reflect the three dimensions of engagement: (i) vigor; (ii) absorption; and (iii) dedication, each dimension is represented by three items that will be evaluated through a Likert-type scale, ranging from "never" (0 points) to "always" (6 points).
Learning perception | 6 months
  Learning perception in mathematics and in general studies will be assessed by means of a questionnaire consisting of eight items. Items 1- 4 will assess the "perceived learning" dimension and items 5-8 will measure the "satisfaction with learning" dimension. All items will be scored according to a five-point Likert scale, where "1" is (strongly disagree) and "5" is (strongly agree).
Academic performance | 6 months
  Academic performance will be evaluated through the marks reported by the schools before and after the intervention.
Inhibition | 6 months
  Inhibition will be evaluated through the Flanker task protocol, part of the NIH Examiner programme. This is a computerised programme where the subject answers the tests individually. The algorithm provided by the program, ranging from 0 to 10, which includes accuracy and reaction time, will be recorded.
Cognitive flexibility | 6 months
  Cognitive flexibility will be evaluated through the Shifting task protocol, part of the NIH Examiner programme. This is a computerised programme where the subject answers the tests individually. The algorithm provided by the program, ranging from 0 to 10, which includes accuracy and reaction time, will be recorded.
Working memory | 6 months
  Working memory will be evaluated through the N-Back protocol, part of the NIH Examiner programme. This is a computerised programme where the subject answers the tests individually. The algorithm provided by the program, ranging from 0 to 10, which includes accuracy and reaction time, will be recorded.
Novelty | 6 months
  Novelty will be assessed through the Novelty Need Satisfaction Scale. Five of the 19 questions that make up the original scale will be selected and participants will be asked to answer them on a Likert-type scale where 1 = "strongly disagree" and 5 = "strongly agree".
School climate | 6 months
  School climate will be assessed using the students' perception of school climate scale (PACE-33). Fifteen items will be evaluated. All items will be scored according to a five-point Likert scale, where "1" is (strongly disagree) and "5" is (strongly agree).
Enjoyment and boredom | 6 months
  Enjoyment and boredom will be assessed using the Spanish version of The Sport Satisfaction Instrument. This scale is composed of eight items. Participants will have to rate their degree of agreement with the items referring to fun or boredom on a five-point Likert-type scale, ranging from 1 (strongly disagree) to 5 (strongly agree).
Dietary patterns | 6 months
  Adherence to the Mediterranean diet will be measured using the updated version 2.0 of the KIDMED questionnaire.
Sociodemographic characteristics | 6 months
  Sociodemographic characteristics will be measured through the Spanish-adapted version III of The Family Affluence Scale. This scale is composed of six questions . Each question is scored on a categorical scale, and the sum of the scores from the six items result in an aggregate index ranging from 0 to 13.
Teachers' perceptions about the feasibility of the intervention program. | 6 months
  Perception about the suitability and the development of the intervention program (perceptions, barriers, points to improve, strengths...) a semi-structured interview will be conducted with the teachers involved in the intervention.
Students' perceptions about the feasibility of the intervention program. | 6 months
  A discussion group will be developed for each of the proposed interventions with a subsample of students, in order to obtain information on the suitability and development of the intervention programme (perceptions, barriers, areas for improvement, strengths, etc.).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Extremadura, Cáceres, Spain

REFERENCES:
- [Derived] Grao-Cruces A, Martin-Acosta F, Vaquero-Solis M, Ruiz-Hermosa A, Camiletti-Moiron D, Sanchez-Oliva D. Fitness, Weight Status and Executive Functions in Adolescents: A Cluster Analysis. Scand J Med Sci Sports. 2025 Aug;35(8):e70098. doi: 10.1111/sms.70098. PMID 40719569
- [Derived] Bandera-Campos FJ, Grao-Cruces A, Camiletti-Moiron D, Martin-Acosta F, Munoz-Gonzalez R, Gonzalez-Perez M, Ruiz-Hermosa A, Vaquero-Solis M, Padilla-Moledo C, Sanchez-Oliva D. Effectiveness of a multicomponent intervention to promote physical activity during the school day: rationale and methods of the MOVESCHOOL study. Front Public Health. 2025 Mar 12;13:1565914. doi: 10.3389/fpubh.2025.1565914. eCollection 2025. PMID 40144996